CLINICAL TRIAL: NCT06733883
Title: "I've Got the Music in Me." Music Therapy for Adolescents with Emotional Difficulties: a Clinical Study
Brief Title: Music Therapy for Adolescents with Emotional Difficulties
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Academy of Music (Other)
Responsible Party: Principal Investigator, Anne Margrethe Myhre, Professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 571344
Record Dates: First submitted 2024-01-08; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-01

CONDITIONS: Depressive Disorder; Emotional Dysregulation
Keywords: Music therapy; Adolescents; Emotional dysregulation; Depression
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Psychotherapy

STUDY DESIGN:
Intervention Model Description: Music therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Music therapy (Experimental): All participants get 10 sessions of music therapy, each lasting for 45 to 60 minutes.
  Interventions: Other: psychotherapy

INTERVENTIONS:
Other: psychotherapy — Music therapy

SUMMARY:
The goal of this clinical trial is to examine the effects of a music therapy program in adolescents aged 13-18 years old with emotional difficulties, primarily depression and possibly concurrent diagnoses of anxiety.

The main questions are:

* What recruitment methods, barriers, and facilitators influence study participation among adolescents with emotional difficulties receiving music therapy in the present study?
* Does music therapy contribute to a significant reduction in depression and anxiety symptoms, inclusive concomitant symptoms?
* How do adolescents with emotional disorders perceive participation in music therapy, and how do they articulate its potential impacts on their health and well-being?

Participants will be invited to participate in a music therapy program, in addition to standard treatment given (TAU). They meet individually in the clinic with a professional music therapist once a week over a period of ten weeks. They will also do musical home exercises between the sessions. Psychiatric interviews and clinical assessments will be conducted before treatment. Assessments and questionnaires will be performed right after the therapy program and three months after ended therapy. There will also be conducted qualitative interviews with a subgroup of the participants.

DETAILED DESCRIPTION:
Background Globally, emotional distress encompassing depression and anxiety is recognized as a predominant contributor to illness and disability among adolescents. These disorders substantially reduce adolescents' quality of life and account for a significant portion of disability-adjusted life years (DALYs). Existing treatment, which typically includes various forms of psychotherapy, possibly augmented with psychopharmaca, demonstrate only moderate efficacy. In Norway, over half of adolescents referred to specialized mental health services have depressive symptoms or ideation as their reason for referral. A substantial fraction of this population is diagnosed with depression either as the main condition or co-morbid with anxiety or other emotional difficulties.

Empirical evidence from a series of controlled intervention studies underscores the beneficial effects of music therapy on adults with depressive disorders, resulting in significant symptom alleviation and improved daily functionality. Additionally, research focusing on the impact of music therapy for adults with anxiety has demonstrated a significant reduction in symptoms.

However, research into the potential efficacy of music therapy for adolescents suffering from depression and anxiety remains relatively sparse. Preliminary studies indicate that music therapy may serve as a valuable intervention, reducing symptoms associated with these conditions. Nevertheless, existing research exhibits considerable variation in populations, methodologies, study designs, and outcome assessments. Furthermore, these studies incorporate both active and passive music therapy techniques, complicating the determination of optimal methodological approaches. Moreover, none of these studies have examined the supplementary benefits of integrating music therapy with standard treatment protocols for adolescents' depression, such as cognitive behavioral therapy (CBT) and pharmacotherapy.

Additionally, incidents of self-harm and suicidal ideation remain unreported in these studies. The present study aims to address these gaps in the existing literature and evaluate the potential applicability of positive outcomes observed in adult music therapy to adolescents with emotional disorders such as depression and anxiety.

A preliminary pilot study was conducted between autumn 2021 and June 2022, including five adolescents aged 13 - 18 years. This pilot study was designed to evaluate the recruitment and music therapy procedure for a larger-scale study. Among the three who completed the study, a significant reduction in depressive symptoms was observed from pre- to post-intervention. The participants reported enhanced coping mechanisms post-intervention, appreciating the therapeutic "time out" from challenging emotions and thoughts. Self-reports from the participants and feedback from therapists, indicated improved daily functioning during the music therapy intervention period.

Considering the reviewed literature and the findings from the pilot study, the following research questions will be explored:

1. What recruitment methods, barriers, and facilitators influence study participation among adolescents with emotional difficulties receiving music therapy in the present study?
2. Does music therapy contribute to a significant reduction in depression and anxiety symptoms, including concomitant symptoms?
3. How do adolescents with emotional disorders perceive participation in music therapy, and how do they articulate its potential impacts on their health and well-being?

Method

The study employs a single-arm repeated measures design, integrating both quantitative and qualitative data collection methods. It is conducted in collaboration between The Norwegian Academy of Music and Oslo University Hospital (OUH) and has received approval from the Regional Ethical Committee (REC) and the Patient Protection Representative at OUH.

20 adolescents aged 13 to 18 years, diagnosed with emotional disorders such as depression and/or anxiety, will be recruited from a child and adolescent outpatient unit in eastern Norway. They will receive standard treatment, including cognitive therapy potentially supplemented with psychopharmacological interventions, in addition to music therapy.

Participants will be referred to the study via two potential pathways. First, participants already receiving treatment at the clinic, who may require supplementary interventions to verbal therapy, may be referred by their current therapist to the music therapist. Alternatively, team leaders will identify new patients suitable for the study. Based on the diagnostic assessments, adolescents diagnosed with depressive episodes, anxiety, or in combination with other psychiatric disorders will be invited to supplement their standard treatment with music therapy. Exclusion criteria include diagnoses of autism spectrum disorders or intellectual disabilities, as well as severe depressive episodes and high suicidal risk, given that these conditions require more intensive care.

The music therapy program comprises ten weekly individual sessions. The initial session will include an introductory conversation to assess participants' musical preferences, resources, and history. Each session will last 45 to 60 minutes and will include warm-up exercises involving stretching, vocalization, and breathing techniques, followed by active music therapy with reproduction of popular music. Sessions will conclude with music listening and creation of a playlist for home listening. The therapy will be based on relational, humanistic and resource-oriented approaches to music therapy.

Prior to inclusion in the study, potential participants will be screened by a specialist in child and adolescent psychiatry using KIDDIE-SADS (Schedule for Affective Disorders and Schizophrenia) to ensure appropriateness and accuracy of their diagnoses for the study.

Data will be collected at three time points: at baseline, within one week following the completion of the music therapy, and at follow-up three months later.

The quantitative assessment will utilize the following measures:

* Beck's Depression Inventory (BDI-II) to assess depressive symptoms.
* The Multidimensional Anxiety Scale for Children (MASC) to evaluate anxiety symptoms.
* The Inventory of Life Quality (ILC) to measure quality of life.
* The Suicidal Ideation Questionnaire (SIQ-JR) to assess suicidal ideation.
* The Self-Harm Inventory (SHI) to assess self-harm behaviors.
* The Difficulties in Emotion Regulation Scale (DERS) to measure difficulties in emotional regulation.
* The Healthy-Unhealthy Music Scale (HUMS) to investigate the relationship between music and emotional experiences.

The qualitative assessment will utilize the following methods:

All participants will be interviewed within one week after the music therapy intervention is concluded, and at follow-up three months later. During the interviews, conducted by the music therapist, participants will be encouraged to provide feedback on the music therapy program, suggest improvements, and reflect on the therapy's impact on their health and behavior. These insights will contribute to the development of hypotheses and models to understand the mechanisms by which music therapy benefits this population and enhance well-being.

These interviews will be subjected to an inductive thematic analysis, where the goal is to gain deeper insight into the participants' experiences with the music therapy program.

Results

The findings of the study will be disseminated through publications in international peer-reviewed journals.

Ethics

Several ethical aspects, such as informed consent, confidentiality, and the protection of participant data, require careful consideration. Informed consent will be obtained through specifically designed forms; one for the participants aged 16 and above, who can provide their own consent, and another for the parents of participants under 16.

It is imperative to communicate to all participants their right to withdraw from the study at any stage, including during the course. All data and sensitive information must be securely stored in locked cabinets. Record-keeping will be conducted using an electronic journal system for Norwegian hospitals (DIPS), the computer system employed by the child and adolescent outpatient unit, while collected data will be stored in MedInsight and coded to ensure confidentiality. The balance between potential benefits and harms must be carefully considered when involving children in research, particularly in relation to the research theme. In this study, participants will engage in music activities and conversations, designed to promote mastery, curiosity, and highlight the participants' resourses. The research has the potential to benefit children and young people receiving treatment at the child and adolescent's outpatient unit, should the findings support the recommendation of music therapy as a treatment option.

The study will guarantee a safe environment for all participants. A crisis management plan outlining procedures to be followed if a participant expresses intent to harm themselves or others, will be established. Continuous collaboration with the responsible practitioner will be maintained throughout the data collection.

ELIGIBILITY:
Inclusion criteria:

* adolescents 13 to 18 years
* emotional difficulties

Exclusion criteria:

* autism spectrum disorder
* mental retardation
* severe depressive episode combined with high suicidal risk

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Beck's Depression Inventory | The inventory will be assessed at three time points: at baseline, one week post-intervention, and three months post-intervention
  The inventory is a 21-item self-report instrument used to measure the severity of depression. The minimum score is zero, indicating no symptoms or signs of depression, while the maximum score is 63, indicating severe depression.
The Satisfaction Scale | The scale will be used at two time points: one week post-intervention, three months, post-intervention
  Participants provide feedback on their experience with participating in the study by indicating their level of agreement with six statements, rated on a scale from 1 to 5, where 1 signifies 'strongly disagree' and 5 signifies 'strongly agree' (see attached questionnaire). The minimum score is six, indicating no satisfaction, while the maximum score is 30, indicating high degree of satisfaction.

SECONDARY OUTCOMES:
Spence Children's Anxiety Scale | The scale will be used at three time points: at baseline, one week post-intervention, and three months post-intervention
  The Scale is a 45-item self-report questionnaire that covers a broad range of anxiety symptoms in children and adolescents. Minimum score is zero which means no symptoms or signs of anxiety. Maximum score is 114 which indicate severe anxiety.
Inventory of Life Quality in Children and Adolescents | The inventory will be assessed at three time points: at baseline, one week post-intervention, and three months post-intervention.
  The inventory is a 7-item assessment tool administered as a self-report questionnaire. It is designed to evaluate the quality of life in young individuals. This inventory is utilized to measure various dimensions of life satisfaction and well-being in children and adolescents, covering both physical and psychosocial aspects. Responses to items are rated on a Likert-type scale, where respondents indicate the frequency or intensity of their experiences. 1 = Never/Not at all. 5 = Always/Extremely. The minimum possible score is 7, indicating very poor quality of life across all assessed domains. The maximum total score 35, indicating excellent quality of life across all assessed domains.
Suicidal Ideation Questionnaire | The questionnaire will be used at three time points: at baseline, one week post-intervention, and three months post-intervention
  The Questionnaire is a 15-item self-report questionnaire designed to measure the frequency and intensity of suicidal thoughts in individuals, particularly adolescents. The questionnaire is used to identify individuals who may be at risk for suicidal behavior. The questionnaire is scored on a Likert-type scale, where each item is rated from 0 ("I never had this thought") to 6 ("This thought was almost always on my mind"). The individual scores for each item are summed to obtain a total score. The minimum possible score is zero, indicating no suicidal thoughts at any time during the specified period. The maximum score is 90, indicating high frequency and intensity of suicidal ideation in the specified period.
Deliberate Self-Harm Inventory | The inventory will be assessed at three time points: baseline, one week post-intervention, and three months post-intervention
  The inventory is a structured 17-item assessment tool designed to measure the occurrence and characteristics of deliberate self-harm behaviors in individuals. This inventory is commonly used in both clinical and research settings to assess self-injurious actions that are intentionally performed, without suicidal intent, for various psychological reasons. The minimum score is zero, indicating that the individual has not engaged in any form of deliberate self-harm.
  The maximum score is 17, indicating engagement in all the types of self-harming behaviors listed.
Difficulties in Emotion Regulation Scale | The scale will be used at three time points: at baseline, one week post-intervention, and three months post-intervention
  The Scale consists of 36 items, each rated on a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always). It is a comprehensive self-report instrument designed to assess emotional dysregulation across multiple dimensions. This scale is widely used to evaluate how individuals experience and manage their emotions. It is particularly useful in understanding the emotional regulation challenges that are central to various psychological disorders.
  The minimum score is 36, which would indicate no difficulties in emotion regulation. The maximum score is 180, indicating severe difficulties in emotion regulation.
Healthy-Unhealthy Music Scale | The scale will be used at three time points: at baseline, one week post-intervention, and three months post-intervention
  The scale is a 13-item assessment tool administered as a self-report questionnaire. It is designed to evaluate individuals' listening habits and preferences regarding music, and how these habits potentially influence their emotional and psychological well-being. This scale is used primarily to understand the role of music in mental health, specifically looking at the dichotomy between healthy and unhealthy music engagement. The items are rated on a Likert-type scale, ranging from 1 to 5, where a higher score represents a stronger agreement or preference. The Healthy Music Engagement Subscale consists of 5 items summing the scores of items related to healthy music use. The minimum score is 5, indicating minimal engagement with music, and the maximum score is 25 indicating maximal engagement with music. The Unhealthy Music Engagement Subscale consists of 8 items summing the scores of items related to unhealthy music use.

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Myhre, MD Phd, Principal Investigator — Oslo UH
Locations (1):
- Oslo university hospital, Oslo, Nydalen, Norway

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in the publication of the Phd will be shared within the reseach-group after they are deidentified. A coding list is available for the PI in the study. The Phd student can also see and add participants to the study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will become available from start of the inclusion to the study is completed.
Access Criteria: The PI is responsible for the data. Members of the reseachgroup have access to the data and are approved by the Regional Ethical Committee.

REFERENCES:
- [Background] Aasen, H. (2001). An empirical investigation of depression symptoms: norms, psychometric characteristics, and factor structure of the Beck Depression Inventory II. Bergen: Det psykologiske fakultet, Universitetet i Bergen.
- [Background] Aalbers S, Fusar-Poli L, Freeman RE, Spreen M, Ket JC, Vink AC, Maratos A, Crawford M, Chen XJ, Gold C. Music therapy for depression. Cochrane Database Syst Rev. 2017 Nov 16;11(11):CD004517. doi: 10.1002/14651858.CD004517.pub3. PMID 29144545
- [Background] Bakken, A. & Osnes, S.M. (2021). Ung i Oslo 2021. Ungdomsskolen og videregående skole. NOVA Rapport 9121. Oslo: NOVA, OsloMet
- [Background] Belski N, Abdul-Rahman Z, Youn E, Balasundaram V, Diep D. Review: The effectiveness of musical therapy in improving depression and anxiety symptoms among children and adolescents - a systematic review. Child Adolesc Ment Health. 2022 Nov;27(4):369-377. doi: 10.1111/camh.12526. Epub 2021 Dec 1. PMID 34854208
- [Background] Erkkila J, Brabant O, Hartmann M, Mavrolampados A, Ala-Ruona E, Snape N, Saarikallio S, Gold C. Music Therapy for Depression Enhanced With Listening Homework and Slow Paced Breathing: A Randomised Controlled Trial. Front Psychol. 2021 Feb 16;12:613821. doi: 10.3389/fpsyg.2021.613821. eCollection 2021. PMID 33664693
- [Background] FHI. (2015, 11.05). Fakta om sosial støtte og ensomhet. Hentet 07.04 2020 fra https://www.fhi.no/fp/psykiskhelse/psykiskelidelser/sosial-stotte-og-ensomhet--- faktaar/ FHI. (2018, 14.05).
- [Background] Gross, J. J. (2013). Emotion Regulation: Conceptual Foundations. In J. J. Gross (Ed.), Handbook of Emotion Regulation, Second Edition (Second edition. ed., pp. 3-22): Guilford Publications.
- [Background] Grøholt B og Sund AM. (2019). Depressive lidelser. Veileder i barne- og ungdomspsykiatri. Den norske legeforeningen
- [Background] Geretsegger M, Mossler KA, Bieleninik L, Chen XJ, Heldal TO, Gold C. Music therapy for people with schizophrenia and schizophrenia-like disorders. Cochrane Database Syst Rev. 2017 May 29;5(5):CD004025. doi: 10.1002/14651858.CD004025.pub4. PMID 28553702
- [Background] Hendricks CB, Robinson B, Bradley B, et al. (1999). Using music techniques to treat adolescent depression. J. Humanist. Couns. Educ Dev. 38: 39-46.
- [Background] Helsedirektoratet (2013). Nasjonal faglig retningslinje for utredning, behandling og oppfølging av personer med psykoselidelser.
- [Background] Ishak M, Herrera N, Martin C, et al.(2021). Music Therapy for Depression in Adolescents: A Systematic Review of Randomized Controlled Trials. Int J Psychiatr Res. 2021; 4(1): 1-5.
- [Background] Johns, U. (2008). " Å bruke tiden - hva betyr egentlig det?" Tid og relasjon - et intersubjektivt perspektiv. NMH-publikasjoner; 2008:3. Skriftserie fra Senter for musikk og helse;1. Norges musikkhøgskole
- [Background] Jozefiak T, Larsson B, Wichstrom L. Changes in quality of life among Norwegian school children: a six-month follow-up study. Health Qual Life Outcomes. 2009 Feb 4;7:7. doi: 10.1186/1477-7525-7-7. PMID 19193211
- [Background] Kaufman J, Birmaher B, Axelson D, Pereplitchikova F, Brent D, Ryan N. (2016). The KSADS-PL DSM-5. Kennedy Krieger Institute. Baltimore.
- [Background] Monsen, J. T., Solbakken, O. A. (2013). Affektintegrasjon og nivåer av mental representasjon: Fokus for terapeutisk intervensjon i Affektbevissthetsmodellen. Tidsskrift for norsk psykologforening, 50, 8, 740-752.
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Norsk pasientregister (NPR) 2019. Helsedirektoratet.
- [Background] Porter ME, Larsson S, Lee TH. Standardizing Patient Outcomes Measurement. N Engl J Med. 2016 Feb 11;374(6):504-6. doi: 10.1056/NEJMp1511701. No abstract available. PMID 26863351
- [Background] Reynolds R (1987). Suicidal Ideation Questionnaire: Professional manual. Psychological Assessment Resources Inc.
- [Background] Rolvsjord, R. (2010). Resource oriented music therapy in mental health care. Barcelona Publishers.
- [Background] Ruud, E. (2008). Et humanistisk perspektiv på musikkterapi. Norges musikkhøgskole Skriftserie fra Senter for musikk og helse;1. NMH-publikasjoner;2008:3
- [Background] Ruud, E. (2020) Towards a Sociology of music therapy: Musicking as a cultural Immunogen. Barcelona publishers.
- [Background] Sansone RA, Sansone LA. Measuring self-harm behavior with the self-harm inventory. Psychiatry (Edgmont). 2010 Apr;7(4):16-20. PMID 20508804
- [Background] Trondalen, G. (2016). Relational Music Therapy: An Intersubjective Perspective. Dallas, TX: Barcelona Publishers.
- [Background] WHO (2005). Promoting Mental Health, Concepts; Emerging EvidencePractice. A Report of the World Health Organization, Department of Mental Health and Substance Abuse in collaboration with the Victorian Health Promotion Foundation and The University of Melbourne.
- [Background] Saarikallio S, Gold C, McFerran K. Development and validation of the Healthy-Unhealthy Music Scale. Child Adolesc Ment Health. 2015 Nov;20(4):210-217. doi: 10.1111/camh.12109. Epub 2015 May 18. PMID 26726295
- [Background] Bellapu, A., Chemmanoor, S., Hu, M., Kim, N., & Clark, C. (2021). Journal of Student Research, 10(4). https://doi.org/10.47611/jsrhs.v10i4.2385)